CLINICAL TRIAL: NCT04662437
Title: The Status of Parathyroid Hormone Secretion and Its Relationship With White Blood Cells, Neutrophil / Lymphocyte Ratio, c Reactive Protein, Fibrinogen, Procalcitonin, Ferritin and D-dimer in Hospitalized Covid-19 Patients
Brief Title: The Status of Parathyroid Hormone Secretion in Covid-19 Patients
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Didem Ertorul (Unknown)
Responsible Party: Principal Investigator, Sabahattin Destek, Associate Professor, Bezmialem Vakif University
Other Study IDs: 08122020
Record Dates: First submitted 2020-12-08; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: COVID-19 Infection; Parathyroid Gland; Parathyroid Hormone; Calcium; Phosphorus; Alkaline Phosphatase
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 Patient Group: 10 ml of venous blood was taken from the forearm venous vein from people in the Covid-19 Patient Group, and the level of parathyroid hormone, calcium, phosphorus, alkaline phosphatase was measured from this blood.
  Interventions: Diagnostic Test: Venous blood was collected for biochemistry testing
- Healthy Control Group: 10 ml of venous blood will be taken from the forearm venous vein from the healthy control group and the parathyroid hormone, calcium, phosphorus, alkaline phosphatase level will be measured from this blood.
  Interventions: Diagnostic Test: Venous blood was collected for biochemistry testing

INTERVENTIONS:
Diagnostic Test: Venous blood was collected for biochemistry testing — From the people in the healthy control group, 10 ml of venous blood was collected from the venous vein in the forearm of all individuals in the study. Parathyroid hormone, calcium, phosphorus, alkaline phosphatase levels were measured from this blood.

SUMMARY:
COVID-19 infection causes a hypersensitive immune reaction and widespread inflammation in various organs of the body, especially through cytokines in the lungs. This cytokine-mediated widespread inflammation can also affect the parathyroid glands, resulting in impaired parathyroid secretion.

Researchers evaluated the levels of parathyroid hormone, calcium, phosphorus, and alkaline phosphatase in patients hospitalized for COVID-19 infection. Researchers excluded patients on intensive care therapy and patients with known parathyroid disease.

The researchers examined the association of parathyroid hormone secretion with COVID-19 disease, white blood cells, neutrophil / lymphocyte ratio, C reactive protein, fibrinogen, procalcitonin, ferritin, and D-dimer in these patients. The researchers compared the parathyroid hormone level of healthy people without COVID-19 infection and known parathyroid disease with the parathyroid hormone level of Covid-19 patients.

DETAILED DESCRIPTION:
The coronavirus-2 (SARS-COV-2) virus, which can cause severe acute respiratory syndrome through the droplet, has caused the global Coronavirus 19 (COVID-19) pandemic. COVID-19 infection can be asymptomatic or lead to serious illness and even death. This virus causes a hypersensitive immune reaction and varying degrees of widespread inflammation through cytokines in various organs of the body, mainly the lungs.

Cytokine-mediated widespread inflammation caused by the virus may also affect the parathyroid glands, causing their functions to deteriorate. Thus, it may cause changes in parathyroid hormone secretion.

The researchers evaluated the results of serum parathyroid hormone, calcium, phosphorus, alkaline phosphatase tests in patients who were symptomatic and hospitalized with COVID-19 infection. Participants also evaluated the relationship of parathormone with white blood cells, neutrophil / lymphocyte ratio, c reactive protein, fibrinogen, procalcitonin, ferritin, and D-dimer in these patients. The researchers compared the parathyroid hormone levels of patients with COVID-19 infection with the parathyroid hormone levels of healthy individuals without COVID-19 infection and parathyroid disease. So the investigators looked for differences in parathyroid hormone levels between both groups. Researchers did not include patients in the intensive care unit and patients with known parathyroid disease.

ELIGIBILITY:
Inclusion Criteria:

* To accept research.
* Being over the age of 18.
* COVID 19 test results to be positive.
* Not taking parathyroid disease medication before.
* Receiving inpatient treatment in the COVID service in the hospital.

Exclusion Criteria:

* Not accepting research.
* Be under the age of 18.
* Negative COVID 19 test results for patients.
* COVID patients treated as outpatient.
* Parathyroid disease in the healthy control group.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalized and treated for COVID-19 without parathyroid disease were formed.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Comparison of parathyroid hormone between groups | 90 days
  In the study, serum parathyroid hormone results of the Covid patient group and non-Covid control groups were recorded and compared statistically.
Comparison of calcium between groups | 90 days
  In the study, serum calcium results of the Covid patient group and non-Covid control groups were recorded and compared statistically.
Comparison of phosphorus between groups | 90 days
  In the study, serum phosphorus results of the Covid patient group and non-Covid control groups were recorded and compared statistically.
Comparison of alkaline phosphatase between groups | 90 days
  In the study, serum alkaline phosphatase results of the Covid patient group and non-Covid control groups were recorded and compared statistically.
White blood cells (WBC) results of Covid 19 patient group | 90 days
  In the study, serum WBC results were recorded in Covid 19 patient groups.
Neutrophil / lymphocyte ratio (N/LO) results of Covid 19 patient group | 90 days
  In the study, serum N/LO results were recorded in Covid 19 patient groups.
C-reactive protein (CRP) results of Covid 19 patient group | 90 days
  In the study, serum CRP results were recorded in Covid 19 patient groups.
Fibrinogen results of Covid 19 patient group | 90 days
  In the study, serum fibrinogen results were recorded in Covid 19 patient groups.
Procalcitonin results of Covid 19 patient group | 90 days
  In the study, serum procalcitonin results were recorded in Covid 19 patient groups.
Ferritin results of Covid 19 patient group | 90 days
  In the study, serum ferritin results were recorded in Covid 19 patient groups.
D-dimer results of Covid 19 patient group | 90 days
  In the study, serum D-dimer results were recorded in Covid 19 patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Özalp Çelikçi, Dr, Study Chair — Sancaktepe Education and Research Hospital
Locations (1):
- Bezmialem VU, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study will be shared when it becomes an article.

REFERENCES:
- [Result] Sun JK, Zhang WH, Zou L, Liu Y, Li JJ, Kan XH, Dai L, Shi QK, Yuan ST, Yu WK, Xu HY, Gu W, Qi JW. Serum calcium as a biomarker of clinical severity and prognosis in patients with coronavirus disease 2019. Aging (Albany NY). 2020 Jun 25;12(12):11287-11295. doi: 10.18632/aging.103526. Epub 2020 Jun 25. PMID 32589164
- [Result] di Filippo L, Formenti AM, Doga M, Frara S, Rovere-Querini P, Bosi E, Carlucci M, Giustina A. Hypocalcemia is a distinctive biochemical feature of hospitalized COVID-19 patients. Endocrine. 2021 Jan;71(1):9-13. doi: 10.1007/s12020-020-02541-9. Epub 2020 Nov 9. No abstract available. PMID 33165763
- [Result] Somasundaram NP, Ranathunga I, Ratnasamy V, Wijewickrama PSA, Dissanayake HA, Yogendranathan N, Gamage KKK, de Silva NL, Sumanatilleke M, Katulanda P, Grossman AB. The Impact of SARS-Cov-2 Virus Infection on the Endocrine System. J Endocr Soc. 2020 Jul 2;4(8):bvaa082. doi: 10.1210/jendso/bvaa082. eCollection 2020 Aug 1. PMID 32728654